CLINICAL TRIAL: NCT05879952
Title: Virtual Reality and Neuropsychiatric Rehabilitation: a Single-blind, Randomized, Controlled Pilot Study in Patients With Global Developmental Delay.
Brief Title: Virtual Reality and Neuropsychiatric Rehabilitation in Patients With Global Developmental Delay.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesca Cucinotta, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nir01
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Global Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The group consists of 50 patients diagnosed with global developmental delay, randomply assigned.
  The patients underwent treatment as usual (TAU) integrated with the use of BTsN pediatric modules, in a 1:1 ratio. All the exercises have been customized by the therapists according to the individual treatment needs, adapting the level of difficulty to the patient's abilities.
  Overall, each patient was treated over a period of 6 months, up to a total of n. 48 sessions, twice a week, lasting 45 minutes each.
  Interventions: Behavioral: TAU + BTsN session
- Control Group (CG) (Active Comparator): The group consists of 50 patients diagnosed with global developmental delay randomply assigned.
  The patients underwent TAU, consisting in standard neuro-psychomotor training. The treatment was tailored according to each child's goals need and preferences.
  Overall, each patient was treated over a period of 6 months, up to a total of n. 48 sessions, twice a week, lasting 45 minutes each.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TAU + BTsN session — BTsN treatment session included exercises aimed at identifying, finding, chasing or moving objects, with the aim of improving the perceptual-cognitive skills of each patient, through audio-visual stimuli and feedback implementing visuo-spatial skills and spatial cognition, allowing at the same time motor coordination and balance improvement.
  Other Names: standard neuro-psychomotor training + virtual reality game sessions
  Arms: Experimental Group (EG)
Behavioral: TAU — neuro-psychomotor training promotes a better organization of global motor skills, improve hand-eye coordination, promote the development of language as communication, enriching representation and symbolization skills.
  Other Names: neuro-psychomotor training
  Arms: Control Group (CG)

SUMMARY:
Global Developmental Delay is a disorder characterized by failure achievement of expected milestones in different areas of psychomotor development before 5 years of age. Recent data in the literature have emphasized the importance of early therapeutic intervention. However, few specific interventions have been described in the literature for this disorder.

Among the high-tech tools used in recent years for rehabilitation, the BTs Nirvana is one of the semi-immersive system that can also be used in children, which allows to stimulate cognitive and motor domains. Objective of this single-blind, randomized, controlled study is to evaluate the feasibility and the effectiveness of integrated rehabilitation treatments with the use of BTs Nirvana in patient with Global Developmental Delay.

DETAILED DESCRIPTION:
Global Developmental Delay (GDD) is a disorder characterized by failure achievement of expected milestones in different areas of psychomotor development before 5 years of age. The estimated incidence of GDD is 1-3%, an early diagnosis and an efficacy treatment could provide a better long-term prognosis. Recent literature data have underlined the importance of early diagnosis followed by appropriate therapeutic management. In fact, GDDs could evolve into different neurodevelopmental disorders, especially if associated with other risk factors, such as intrauterine growth retardation, nutrient deficiencies, breastfeeding and maternal education, scarce social and economic conditions, poor learning opportunities, inadequate quality of caregiver-child interactions.

In recent decades, the use of virtual reality (VR) for therapeutic reason has become more and more popular for innovative treatments in cognitive-motor domain. Indeed, VR and the interactive playing can motivate children to learn new skills. Among the high-tech tools used in recent years for rehabilitation, the BTs Nirvana (BTsN) is one of the semi-immersive VR that can also be used in children, which allows to stimulate cognitive and motor domains. The aim of this single-blind, randomized, controlled study is to evaluate the feasibility and the effectiveness of integrated rehabilitation treatments with the use of BTsN in patient with Global Developmental Delay.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diagnosis of GDD, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria;
* age between 12 and 66 months;
* patients without significant medical conditions such as epilepsy, significant visual and auditory sensory deficits, traumatic brain injury, or other significant genetic disorders.
* Signed informed consent and the availability of at least one family member to participate in the diagnostic/therapeutic process.

Exclusion Criteria:

* children not aged between 12 and 66 months;
* significant medical conditions such as epilepsy, significant visual and auditory sensory deficits, traumatic brain injury, or significant genetic disorders.
* Informed consent not signed of at least one family member to participate in the diagnostic/therapeutic process.

Ages: 12 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Griffiths-III Mental Development Scale (GMDS-III) | T0 (Baseline) - T1 (6 Months)
  Assessment tool for children from 0 to 72 months and was for performed to assess Global Quotient (GQ)
Clinical Global Impressions (CGI) | T0 (Baseline) - T1 (6 Months)
  Scale that allows to quantify and monitor patients' progress and response to treatment over time, providing a judgment on global improvement.
Protocol adherence | T0 (Baseline) - T1 (6 Months)
  The number of non-delivered treatment sessions will be counted, and the percentage of deviation will be calculated compared to the total number of treatment sessions.

SECONDARY OUTCOMES:
The Child Behavior Checklist (CBCL 1½-5) | T0 (Baseline) - T1 (6 Months)
  This questionnarie is a caregiver report to identifying problem behavior in children.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neurolesi Bonino Pulejo, Messina, Italy

REFERENCES:
- [Background] Srour M, Mazer B, Shevell MI. Analysis of clinical features predicting etiologic yield in the assessment of global developmental delay. Pediatrics. 2006 Jul;118(1):139-45. doi: 10.1542/peds.2005-2702. PMID 16818559
- [Background] Alderman H, Behrman JR, Glewwe P, Fernald L, Walker S. Evidence of Impact of Interventions on Growth and Development during Early and Middle Childhood. In: Bundy DAP, Silva ND, Horton S, Jamison DT, Patton GC, editors. Child and Adolescent Health and Development. 3rd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2017 Nov 20. Chapter 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK525234/ PMID 30212122
- [Background] Thomaidis L, Zantopoulos GZ, Fouzas S, Mantagou L, Bakoula C, Konstantopoulos A. Predictors of severity and outcome of global developmental delay without definitive etiologic yield: a prospective observational study. BMC Pediatr. 2014 Feb 12;14:40. doi: 10.1186/1471-2431-14-40. PMID 24521451
- [Background] Caliendo M, Di Sessa A, D'Alterio E, Frolli A, Verde D, Iacono D, Romano P, Vetri L, Carotenuto M. Efficacy of Neuro-Psychomotor Approach in Children Affected by Autism Spectrum Disorders: A Multicenter Study in Italian Pediatric Population. Brain Sci. 2021 Sep 14;11(9):1210. doi: 10.3390/brainsci11091210. PMID 34573234
- [Background] Fandakova Y, Hartley CA. Mechanisms of learning and plasticity in childhood and adolescence. Dev Cogn Neurosci. 2020 Apr;42:100764. doi: 10.1016/j.dcn.2020.100764. Epub 2020 Jan 30. No abstract available. PMID 32072937
- [Background] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Background] De Luca R, Naro A, Colucci PV, Pranio F, Tardiolo G, Billeri L, Le Cause M, De Domenico C, Portaro S, Rao G, Calabro RS. Improvement of brain functional connectivity in autism spectrum disorder: an exploratory study on the potential use of virtual reality. J Neural Transm (Vienna). 2021 Mar;128(3):371-380. doi: 10.1007/s00702-021-02321-3. Epub 2021 Mar 6. PMID 33677622
- [Background] Harris K, Reid D. The influence of virtual reality play on children's motivation. Can J Occup Ther. 2005 Feb;72(1):21-9. doi: 10.1177/000841740507200107. PMID 15727045
- [Background] Vasudevan P, Suri M. A clinical approach to developmental delay and intellectual disability. Clin Med (Lond). 2017 Dec;17(6):558-561. doi: 10.7861/clinmedicine.17-6-558. PMID 29196358